CLINICAL TRIAL: NCT02961868
Title: PROgression of FIbromuscular LEsions
Brief Title: Cohort Follow-up of Patients With Renal or Craniocervical Fibromuscular Dysplasia
Acronym: PROFILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de Recherche sur l'Hypertension Artérielle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P071241; P071241 (Other: Assistance Publique - Hopitaux de Paris); 2009-A00288-49 (Other: Agence Française de Securite Sanitaire des Produits de Sante); PHRC-08-192 (Other Grant/Funding Number: Direction Generale de l'Offre de Soin)
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Fibromuscular Dysplasia
Keywords: Renal Artery Obstruction; Carotid Artery Diseases; Genetic Association Studies
MeSH Terms: conditions — Fibromuscular Dysplasia; Renal Artery Obstruction; Carotid Artery Diseases | interventions — Blood Specimen Collection; Biomarkers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prospective cohort (Experimental): 3 years follow-up
  Interventions: Other: Abdominal and supra-aortic trunks vascular imaging; Genetic: Blood sampling (genetic); Other: Blood sampling (biomarkers); Other: Urine sampling

INTERVENTIONS:
Other: Abdominal and supra-aortic trunks vascular imaging — Abdominal and supra-aortic trunks vascular imaging (angiography, CT-angiography or MR-angiography) will be performed 3 years after inclusion. This imaging will be compare to initial imaging (which is a part of usual care, not an intervention added by the study) in order to assess FMD progression.
Genetic: Blood sampling (genetic) — A sample of blood will be taken to meet the objective of estimating the rate of genetic polymorphism that may influence disease progression or be associated with complications.
Other: Blood sampling (biomarkers) — A sample of blood will be taken to biomarkers analysis to meet the primary objective of assessing the risk factors for progression of FMD lesions.
Other: Urine sampling — A sample of urine will be taken to biomarkers analysis to meet the primary objective of assessing the risk factors for progression of FMD lesions.

SUMMARY:
PROFILE is a cohort study evaluating the progression of fibromuscular dysplasia lesions. This study is the prospective dimension of ARCADIA registry (ClinicalTrials.gov Identifier: NCT02884141), which aims to document phenotypic and genetic traits in patients with renal and/or cervical artery fibromuscular dysplasia.

DETAILED DESCRIPTION:
Background

Fibromuscular dysplasia (FMD) is a group of nonatherosclerotic, noninflammatory arterial diseases that usually involve renal and carotid arteries. Patients with FMD may present with renovascular hypertension and/or with cerebrovascular symptoms. The prevalence of FMD in hypertensive patients is estimated at 4/1000. Angiographic classification includes the multifocal type, with multiple stenoses and the 'string-of-beads' appearance that is related to medial FMD, and tubular and focal types which are not clearly related to specific histological lesions. FMD may affect one or more vascular beds and progress to more severe stenosis and to renal or cerebrovascular complications. FMD appears to be familial in 10% of cases (OMIM #135580).

Renal artery FMD may progress to more severe stenosis and to renal atrophy, and/or to stenoses affecting more arteries within or outside the renal vasculature. The risk of progression as assessed from available studies was probably overestimated because documentation of progression was obtained from angiography, a procedure which is not routinely undertaken in patients with favourable clinical and biological outcomes. The disease is progressive, however, and literature stated that patients with FMD should undergo yearly duplex ultrasonography to detect progression of disease, restenosis, or loss of kidney volume.

There are very few data on prognosis of patients with symptomatic carotid or vertebral artery FMD. The risk of arterial disease progression over time is unknown. The risk of ischemic stroke ranged from 0 to about 3% per year in the few studies which assessed that issue.

Objectives

The primary objective is to estimate the incidence and risk factors for progression of FMD lesions. This will be assessed by comparison between initial and 3 years abdominal and supra-aortic trunks vascular imaging (angiography, CT-angiography or Magnetic Resonance (MR) angiography), monitoring of downstream consequences development of lesions progression and clinical events.

The secondary objectives are:

* to estimate rate of genetic polymorphism that may influence disease progression or be associated with complications
* to assess the frequency of multi-site FMD (common objective with the ARCADIA study)
* to collect standardized clinical, radiological, and biological data in patients with FMD through a national registry (common objective with the ARCADIA study)
* to organize a clinical, radiological and biological database and a biobank that will constitute a unique resource to initiate further clinical research (common objective with the ARCADIA study).

ELIGIBILITY:
Inclusion Criteria:

* Patient with renal or craniocervical fibromuscular dysplasia diagnosed during the 2 years before inclusion
* The fibromuscular dysplasia is documented by imaging (angiography, CT-angiography, MR-angiography) of less than 2 years and validated by a radiologist investigator
* Patient who understood and signed inform consent form
* Affiliated to the French health insurance system
* Available for a 3 years follow-up

Exclusion Criteria:

* Patient with renal or craniocervical atherosclerosis, or inflammatory vascular disease as dominant pathological features
* Patient with renal or craniocervical arteries dissection or aneurysm without any other evidence of fibromuscular dysplasia
* Patient under 18 or under tutorship
* Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2009-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Progression of fibromuscular dysplasia lesions confirmed by imaging | 3 years

SECONDARY OUTCOMES:
Glomerular filtration rate (GFR) | Inclusion, 3 years
Kidney height | Inclusion, 3 years
Clinical event: revascularization procedure in a lesion site | Through study completion
Clinical event: renal infarction | Through study completion
Clinical event: ischemic stroke | Through study completion
Clinical event: arterial dissection in a lesion site or downstream from a lesion site | Through study completion
Clinical event: aneurysm rupture in a lesion site or downstream from a lesion site | Through study completion
Prevalence of multisite fibromuscular dysplasia confirmed by imaging | Inclusion, 3 years
Single nucleotide polymorphisms | Inclusion
  Assessed by genome-wide association
Plasminogen/plasmin level | Inclusion
Matrix metalloproteinases level | Inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-François Plouin, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (17):
- Cliniques universitaires Saint-Luc, Brussels, Brussels Capital, Belgium
- France (16):
  - CHU de Bordeaux hopital Saint-Andre, Bordeaux, Aquitaine-Limousin-Poitou-Charentes
  - CHU de Clermont-Ferrand hopital Gabriel-Montpied, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - CHU de Grenoble hopital Albert-Michallon, La Tronche, Auvergne-Rhône-Alpes
  - CHU de Nancy institut Louis-Mathieu, Vandeuvre-les-Nancy, Grand Est
  - CHRU de Lille hopital cardiologique, Lille, Hauts-de-France
  - CHRU de Lille hopital Roger-Salengro, Lille, Hauts-de-France
  - CHU de Caen hopital Cote de Nacre, Caen, Normandy
  - CHU de Toulouse hopital Rangueil, Toulouse, Occitanie
  - AP-HM hopital de la Timone, Marseille, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier de Versailles hopital Andre Mignot, Le Chesnay, Île-de-France Region
  - AP-HP hopital Lariboisiere, Paris, Île-de-France Region
  - AP-HP hopital Pitie-Salpetriere, Paris, Île-de-France Region
  - Centre hospitalier Sainte-Anne, Paris, Île-de-France Region
  - Groupe Hospitalier Paris Saint-Joseph, Paris, Île-de-France Region
  - AP-HP hopital Bichat-Claude-Bernard, Paris, Île-de-France Region
  - AP-HP hopital Tenon, Paris, Île-de-France Region